CLINICAL TRIAL: NCT05677425
Title: Temperature Profiles During Laser Activation in Ureteroscopic Lithotripsy - a Prospective Clinical Study
Brief Title: Temperature Profiles During Laser Activation in Ureteroscopic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 550816
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-02

CONDITIONS: Ureteral Stone
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: Patients ≥ 18 years with a ureteral stone (with or without a concomitant renal stone) and an indwelling nephrostomy tube scheduled for URS lithotripsy at the Day Surgery unit at Haukeland University Hospital, can be enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temperature measurement group (Experimental): Temperature measurement in the renal pelvis during ureteroscopic laser stone disintegration. Temperature measurement will be performed using different laser power settings.
  Interventions: Other: Temperature measurement

INTERVENTIONS:
Other: Temperature measurement — Temperature measurement in the renal pelvis during ureteroscopic laser activation.

SUMMARY:
The primary aim of this study is to investigate the temperature profiles in the renal pelvis during ureteroscopic Thulium Fiber Laser activation using different settings. To this end, comparison of peak temperatures during laser activation for different settings is the main aim. Secondary aim is trying to define the duration of safe laser activation until the threshold for heat induced cell injury (43oC) is reach.

Patients ≥ 18 years with a ureteral stone (with or without a concomitant renal stone) and an indwelling nephrostomy tube scheduled for ureteroscopic lithotripsy at the day surgery unit at Haukeland University Hospital, are eligible to enrolment in the study.

Temperature measurements during ureteroscopic laser stone disintegration will be performed. Follow-up is standardised with clinical consultation and low dose CT 3 months post endoscopically.

DETAILED DESCRIPTION:
BACKGROUND: The Holmium:Yttrium-Aluminium-Garnet (Ho:YAG) has been considered the gold-standard laser for ureteroscopy (URS) because of its versatility, with the ability to break all kinds of stones in the urinary tract as well as tumor- and soft tissue ablation. Development of higher power laser technology has allowed the limits of what can be achieved with URS to be set even higher. In comparison to stone fragmentation, techniques such as dusting and pop-corning often implement higher power settings (>20 Watts), and the efficacy associated with different strategies has been the focus of many studies. Intraoperative safety of URS has gained increased attention, particularly with regard to raised temperature levels. Recently, a new Thulium Fiber Laser (TFL) has been introduced. With the advent of the TFL, discussion surrounding high temperatures during lithotripsy and resultant thermal damage have been fueled further. Defining safe margins for laser settings is especially important for the TFL as no consensus exists for what is acceptable during URS. To date, there are no clinical studies investigating intrarenal temperatures during URS laser treatment. Studying temperature profiles during URS laser activation in patients is therefore of critical importance and highly clinically relevant to define the safety of different laser settings and power.

AIMS OF THE STUDY: The primary aim of this study is to investigate the temperature profiles in the renal pelvis during TFL laser activation using different settings. To this end, comparison of peak temperatures during laser activation for different settings is the main aim. Secondary aim is trying to define the duration of safe laser activation until the threshold for heat induced cell injury (43oC) is reach.

THE URETEROSCOPIC PROCEDURE AND TEMPERATURE MEASUREMENTS: The URS procedure is performed in general anaesthesia and all patients will have prophylactic antibiotics prior to surgery start, either according to urine culture or current local regime.

The procedure starts with a cystoscopy followed by semirigid URS when considered appropriate. Balloon dilatation is performed on demand. When reaching the stone, this is flushed back into the renal pelvis for disintegration there if possible. In cases where the stone cannot be flushed back into the renal pelvis, the stone is disintegrated in situ before the endoscope is advanced up to the renal pelvis for temperature measurements. Before laser disintegration, the semirigid ureteroscope is changed for a flexible ureteroscope that is advanced to the renal pelvis directly or over a guide wire that must be removed as soon as the endoscope is in place. An access sheath cannot be used during this study. Room-tempered (23oC), gravitational irrigation fluid at 60 cm height is used throughout the procedure. Manual pumping should be avoided and should in any case not be performed during the temperature measurements.

Under endoscopic vision, a sterilized thermocouple sensor (K-type, same as in the pre-clinical study) is introduced through the nephrostomy tube so that the tip can identified through the side-holes of the nephrostomy tube. The stone is moved to the central renal pelvis for laser disintegration, and a 150μm laser fiber is introduced into the renal pelvis through the working channel of the flexible ureteroscope. At this point the nephrostomy tube is clamped to achieve filling of the renal pelvis and to mimic a normal procedure.

Laser disintegration of the stone is started using the lowest laser setting of 5 Watts continuously for 120 seconds followed by 60 seconds of idling laser. Temperature measurements are maintained continuously during these 180 seconds, with two measurements per second. When the temperature in the renal pelvis has reached base temperature after one series of measurements, the procedure is repeated for the next laser setting. In total, URS lithotripsy are performed for three different settings. If 43oC is reach during laser activation for any of the laser settings, the laser will be stopped immediately and further laser activation with that specific settings will be aborted. Laser activation with subsequent settings will be ready when base temperature is reached.

If stone treatment is not completed at the end of the three series of laser activation and temperature measurements, further stone disintegration will be performed before finishing the URS procedure.

A double J-stent is placed at the end if deemed necessary by the surgeon. The nephrostomy tube is removed when considered appropriate. If a double J-stent is placed after the procedure, this is removed according to standard routine after 1-2 weeks in the outpatient clinic.

FOLLOW-UP: Follow-up with CT is performed at 3 months post endoscopically for all patients to assess stone free status and exclude a ureteral stricture in addition to a clinical consultation.

LASER SETTINGS: The following laser settings will be used in the study:

5 watts of power: 0.5 Joules (J) / 10 Herz (Hz), short pulse 10 watts of power: 0.5 J / 20 Hz, short pulse 20 watts of power: 0.5 J / 40 Hz, short pulse 30 watts of power: 1 J / 30 Hz, short pulse

ETHICAL CONSIDERATION AND APPROVALS: Participation in the study is voluntarily, and the patient can choose to withdraw at any point during the study process. Inclusion in the study will only be done after the consent form is signed.

The study is approved by The National Committees for Research Ethics in Norway (REK-550816). Application for approval by The Data Protection Authorities at Haukeland University Hospital has been sent.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with a ureteral stone (with or without a concomitant renal stone) and an indwelling nephrostomy tube scheduled for URS lithotripsy at the Day Surgery unit at Haukeland University Hospital

Exclusion Criteria:

* Urinary diversion
* Active infection
* Untreated cancer in the upper urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ulvik, Assoc Prof, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AEsoy MS, Juliebo-Jones P, Beisland C, Ulvik O. Temperature Measurements During Flexible Ureteroscopic Laser Lithotripsy: A Prospective Clinical Trial. J Endourol. 2024 Apr;38(4):308-315. doi: 10.1089/end.2023.0660. Epub 2024 Feb 28. PMID 38185920

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temperature Measurement Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temperature Measurement Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 57 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stone size, mm [Mean (Full Range); unit: mm] | 9 [5 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Temperature Profiles
Description: Temperatures during ureteroscopic laser activation using different laser power settings.
Time Frame: During surgery
Measure: Mean (95% Confidence Interval); unit: Degrees Celcius
Arm/Group | Temperature Measurement Group
Number analyzed (Participants) | 10
Degrees Celcius
  Baseline temperature | 32.5 [31.7 to 33.2]
  Tmax 5 W | 35.3 [34.6 to 36.9]
  Tmax 10 W | 37.9 [36.4 to 39.4]
  Tmax 20 W | 40.0 [39.0 to 41.1]

ADVERSE EVENTS:
Time Frame: From study start until 3 months follow-up.
Description: Adverse events are reported according to Clavien-Dindo.
Arm/Group | Temperature Measurement Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temperature Measurement Group (N=10)
Clavien-Dindo 1 and 2 (Renal and urinary disorders) | 3 (3) — Clavien-Dindo 1 and 2 includes minor adverse events, such as UTI and pain treated with antibiotics and painkillers. Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT05677425/Prot_SAP_000.pdf